CLINICAL TRIAL: NCT00410579
Title: Patient Reported Outcomes in Long Term Survivors With Colon and Rectal Cancer
Brief Title: Patient-Reported Outcomes in Long-Term Survivors of Colon and Rectal Cancers
Status: Completed | Type: Observational
Sponsor: NSABP Foundation Inc (Network)
Collaborators: National Cancer Institute (NCI) (NIH); University of California, Los Angeles (Other)
Responsible Party: Norman Wolmark, MD, NSABP Foundation, Inc.
Other Study IDs: NSABP LTS-01; CDR0000494640 (Other: NCI)
Record Dates: First submitted 2006-12-11; First posted 2006-12-13 (Estimated); Last update posted 2010-12-17 (Estimated); Status verified 2010-12

CONDITIONS: Colorectal Cancer; Fatigue; Long-term Effects Secondary to Cancer Therapy in Adults; Pain; Psychosocial Effects of Cancer and Its Treatment
Keywords: pain; fatigue; long-term effects secondary to cancer therapy in adults; psychosocial effects of cancer and its treatment; stage II rectal cancer; stage III rectal cancer; stage II colon cancer; stage III colon cancer; adenocarcinoma of the colon
MeSH Terms: conditions — Colorectal Neoplasms; Fatigue; Pain; Rectal Neoplasms; Colonic Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients treated in NSABP R-02, R-03, C-05, C-06 or C-07: Study population to be interviewed comprises patients who were treated at least 5 years ago for colon or rectal cancer in NSABP trials R-02, R-03, C-05, C-06 or C-07
  Interventions: Other: Telephone interview

INTERVENTIONS:
Other: Telephone interview — Telephone interview to assess generic health status, quality of life, comorbidity, impact of cancer, use of medical services, health rating, pain, fatigue, activities of daily living, demographics, functional well-being(C-06 only), and neurotoxicity (C-07 only)

SUMMARY:
RATIONALE: Learning about quality of life, symptoms, and health behaviors in colorectal cancer survivors may help to determine the long-term effects of colon and rectal cancer treatments and may help to improve the quality of life for future cancer survivors.

PURPOSE: This clinical trial is looking at patient-reported outcomes in long-term survivors of colon and rectal cancers.

DETAILED DESCRIPTION:
OBJECTIVES:

* Characterize 3 separate types of patient-reported outcomes (quality of life [e.g., generic and disease-specific], functional outcomes [e.g., bowel and sexual function and activities of daily living], and clinical symptoms [e.g., pain, fatigue]) in long-term (5+ years) survivors of colon and rectal cancers in a large national sample recruited from five National Surgical Adjuvant Breast and Bowel Project (NSABP) treatment trials.
* Explore the degree to which patient-reported outcomes are impacted by individual characteristics (e.g., specific predisposing factors, enabling resources, and need), by health behaviors (e.g., use of services for cancer-related and non-cancer-related issues), and, when appropriate, by the specific treatments that were received.
* Examine patient-reported outcomes prior to randomization and treatment, 1 year after treatment, and in long-term follow up > 5 years after diagnosis in patients with colon cancer treated with adjuvant chemotherapy on protocols NSABP C-06 or NSABP C-07.

OUTLINE: This is a cohort, single-group, multicenter study.

Patients complete a one-time, computer-assisted telephone interview assessing their overall quality of life (QOL), disease-specific QOL, function and symptoms (including pain and fatigue), use of healthcare services, prevalence and severity of comorbidity, and demographics.

PROJECTED ACCRUAL: A total of 1,167 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Prior diagnosis of colon or rectal cancer
* At least 5 years since participated in 1 of the following clinical trials:

  * NSABP-R-02
  * NSABP-R-03
  * NSABP-C-05
  * NSABP-C-06
  * NSABP-C-07

PATIENT CHARACTERISTICS:

* Able to speak English

PRIOR CONCURRENT THERAPY:

* As per participation requirements of previous NSABP treatment trials

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population to be interviewed comprises patients who were treated at least 5 years ago for colon or rectal cancer in NSABP trials R-02, R-03, C-05, C-06 or C-07
Sampling Method: Non-Probability Sample
Enrollment: 744 (Actual)
Dates: Start 2006-11; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Types of patient-reported outcomes | After all telephone interviews are completed
  Survey battery for quality of life, functional outcomes, and clinical symptoms from patients from all 5 trails
Degree to which patient-reported outcomes are impacted by individual characteristics, health behaviors, and when appropriate specific treatments that were received | After all telephone interviews are completed
  Long Term Mental and Physical Component Scales, EORTC-CR 38, Individual Characteristics and Health Behaviors, treatment information
Comparison of patient-reported outcomes prior to randomization, 1 year after completion of study treatment, and in long-term follow up > 5 years after diagnosis in patients treated in NSABP C-06 or NSABP C-07 trials | After all telephone interviews are completed
  Four generic subscales of FACT-C and the colorectal cancer subscale, total score of symptoms distress scale, SF-12 Vitality subscale and health rating scale; NTX-R

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Study Chair — NSABP Foundation Inc
Locations (200):
- United States (200):
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Evanston Northwestern Healthcare - Evanston Hospital, Evanston, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Clarian Arnett Cancer Care, Lafayette, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Louisville Oncology at Norton Cancer Institute - Louisville, Louisville, Kentucky
  - Ochsner Health Center - Bluebonnet, Baton Rouge, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Suburban Hospital, Bethesda, Maryland
  - Union Hospital Cancer Program at Union Hospital, Elkton MD, Maryland
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Jordan Hospital Club Cancer Center, Plymouth, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Bay Regional Medical Center, Bay City, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Upper Michigan Cancer Center at Marquette General Hospital, Marquette, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Hattiesburg Clinic, PA at Forrest General, Hattiesburg, Mississippi
  - Hematology & Oncology Clinic, Hattiesburg, Mississippi
  - Southeast Missouri Regional Cancer Center at Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Independence Regional Health Center, Independence, Missouri
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - St. Joseph Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Parvin Radiation Oncology, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Midwest Hematology Oncology Group, Incorporated, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - CCOP - Main Line Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - McLeod Regional Medical Center, Florence, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - CCOP - Scott and White Hospital, Temple, Texas
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Center for Cancer Treatment & Prevention at Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Saint Michael's Hospital Cancer Center, Stevens Point, Wisconsin
  - Marshfield Clinic - Wausau Center, Wausau, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin

REFERENCES:
- [Result] Kunitake H, Zheng P, Yothers G, Land SR, Fehrenbacher L, Giguere JK, Wickerham DL, Ganz PA, Ko CY. Routine preventive care and cancer surveillance in long-term survivors of colorectal cancer: results from National Surgical Adjuvant Breast and Bowel Project Protocol LTS-01. J Clin Oncol. 2010 Dec 20;28(36):5274-9. doi: 10.1200/JCO.2010.30.1903. Epub 2010 Nov 15. PMID 21079140
- [Result] Yothers G, Land SR, Ganz PA, et al.: Neurotoxicity (NT) in colon cancer (CC) survivors from NSABP Protocol C-07 comparing 5-FU + leucovorin (FULV) with the same regimen + oxaliplatin (FLOX): preliminary results from NSABP protocol LTS-01. [Abstract] J Clin Oncol 26 (Suppl 15): A-9575, 2008.
- [Derived] Kunitake H, Russell MM, Zheng P, Yothers G, Land SR, Petersen L, Fehrenbacher L, Giguere JK, Wickerham DL, Ko CY, Ganz PA. Quality of life and symptoms in long-term survivors of colorectal cancer: results from NSABP protocol LTS-01. J Cancer Surviv. 2017 Feb;11(1):111-118. doi: 10.1007/s11764-016-0567-y. Epub 2016 Aug 25. PMID 27562475